CLINICAL TRIAL: NCT03461406
Title: A Prospective, Randomized, Active-Controlled, Single-blind, Parallel Group Clinical Trial to Evaluate the Safety and Efficacy of Fibrin Sealant Grifols (FS Grifols) as an Adjunct to Haemostasis During Surgery in Paediatric Subjects
Brief Title: A Study of Safety and Efficacy of Fibrin Sealant Grifols as an Adjunct to Haemostasis During Surgery in Paediatric Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Grifols, S.A. (Industry)
Responsible Party: Sponsor
Organization: Grifols Therapeutics LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IG1405; 2016-004489-24 (EudraCT Number)
Record Dates: First submitted 2018-03-02; First posted 2018-03-12 (Actual); Results first posted 2023-04-07 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Excessive Bleeding During Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fibrin Sealant Grifols (Experimental): Participants topically applied FS Grifols, which consisted of component 1: human fibrinogen (80 mg/mL) and component 2: human thrombin with calcium chloride (500 IU/mL) solutions filled in syringes and assembled on a syringe holder.
  Interventions: Biological: Fibrin Sealant Grifols
- EVICEL (Active Comparator): Participants topically applied EVICEL, which consisted of component 1: Concentrate of human fibrinogen (BAC 2) (55-85 mg/mL) and component 2: human thrombin (800-1200 IU/mL) solutions. The 2 components (BAC2 and thrombin) were mixed and applied topically.
  Interventions: Biological: EVICEL

INTERVENTIONS:
Biological: Fibrin Sealant Grifols — The FE Grifols solution was applied topically via drip or spray application.
  Other Names: FS Grifols
  Arms: Fibrin Sealant Grifols
Biological: EVICEL — The EVICEL solution was applied topically via drip or spray application.
  Arms: EVICEL

SUMMARY:
The objective of the study is to evaluate if FS Grifols is non-inferior to EVICEL® in terms of the percentage of participants achieving hemostasis at the target bleeding site (TBS) by 4 minutes (T4) from the start of treatment application (TStart) with no occurrence of rebleeding until the completion of the surgical closure by layers of the exposed surgical field containing the TBS (TClosure).

DETAILED DESCRIPTION:
This is a prospective, randomized, active-controlled, single-blind, parallel group clinical trial to evaluate the safety and efficacy of FS Grifols as an adjunct to hemostasis during surgery. Approximately 172 pediatric participants will be enrolled and will be randomly allocated in a 1:1 ratio into 1 of 2 treatment groups: FS Grifols or EVICEL. Enrollment will be monitored by surgery type to ensure at least 50% of the surgical procedures are hepatic.

A specific bleeding site will be defined as the TBS when it is determined by the investigator (the surgeon) that control of bleeding by conventional surgical techniques (including suture, ligature, and cautery) is ineffective or impractical and requires an adjunct treatment to achieve hemostasis.

When the TBS is identified, the investigator will record the precise anatomical location of the TBS, rate the intensity of the bleeding at the TBS (Grade 1-4 according to a 5-point validated bleeding severity scale), and record the size of the approximate bleeding surface, (small, medium, and large). For soft tissue surgery only, the investigator will also record the type of soft tissue (ie, fat, muscle, or connective tissue). In this clinical trial, only participants with a TBS with bleeding of Grade 1 (mild) or Grade 2 (moderate) intensity will be enrolled.

This study includes a Screening Visit to determine participant eligibility, a Baseline Visit, the Surgical Procedure (Day 1), and Post-operative assessments at Days 1, 4, and 30. The total duration of a participant's participation in this study is expected to be no longer than 2 months from the Screening Visit to the Post-operative Day 30 Visit.

ELIGIBILITY:
Inclusion Criteria:

Pre-operative:

1. Less than 18 years of age.
2. Requires an elective (non-emergent), open (non-laparoscopic), pelvic, abdominal, or thoracic (non-cardiac) surgical procedure.
3. Participant and/or participant's legal guardian is willing to give permission for the participant to participate in the clinical trial and provide written informed consent for the participant. In addition, assent must be obtained from pediatric participants who possess the intellectual and emotional ability to comprehend the concepts involved in the clinical trial.

   Intra-operative:
4. Presence of an appropriate (as defined in inclusion criterion 5) parenchymous or soft tissue TBS identified intra-operatively by the investigator (the surgeon).
5. TBS has Grade 1 (mild) or Grade 2 (moderate) bleeding intensity according to the investigator's (the surgeon's) judgment. The intensity of the bleeding at the TBS will be rated by the investigator using the 5-point validated bleeding severity scale.

Exclusion Criteria:

Pre-operative:

1. Admitted for trauma surgery.
2. Unwilling to receive blood products.
3. Known history of severe (eg, anaphylactic) reaction to blood products.
4. Known history of intolerance to any of the components of the investigational product (IP).
5. Female participants who are pregnant, breastfeeding or, if of child-bearing potential (ie, adolescent), unwilling to practice a highly effective method of contraception.
6. Previously enrolled in a clinical trial with FS Grifols.
7. Currently participating, or during the study is planned to participate, in any other investigational device or medicinal product study without prior and explicit approval from the sponsor.

   Intra-operative:
8. An appropriate parenchymous or soft tissue TBS (as defined in exclusion criteria 9 and 10) cannot be identified intra-operatively by the investigator (the surgeon).
9. TBS has Grade 3 (severe) bleeding according to the investigator's (the surgeon's) judgment that cannot be controlled with conventional surgical techniques to Grade 1 or Grade 2 bleeding. The intensity of the bleeding at the TBS will be rated by the investigator using the 5-point validated bleeding severity scale.
10. TBS is in an actively infected surgical field.
11. Occurrence of major intra-operative complications that require resuscitation or deviation from the planned surgical procedure.
12. Application of any topical hemostatic agent on the resection surface of parenchyma or soft tissue prior to application of the IP.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 186 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (40):
- United States (12):
  - Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - University of Michigan, Michigan Center, Michigan
  - The Urological Institute of Northeastern New York, Albany, New York
  - Columbia Medical Center, New York, New York
  - St. Christophers Hospital, Philadelphia, Pennsylvania
  - MUSC Health-Children's Hospital, Charleston, South Carolina
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Children's Medical Center Dallas, Dallas, Texas
  - El Paso Childrens Hospital, El Paso, Texas
  - Memorial Hermann Memorial City, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Carilion Children's Pediatric Surgery, Roanoke, Virginia
- Bulgaria (6):
  - MHAT City clinic - Sveti Georgi, Montana
  - UMHAT Dr. Georgi Stranski, Pleven
  - UMHAT Sveti Georgi, Plovdiv
  - UMHAT Kanev, Rousse
  - UMHATEM N.I.Pirogov, Sofia
  - UMHAT Prof. Dr. Stoyan Kirkovich, Stara Zagora
- British Columbia's Children's Hospital, Vancouver, Canada
- France (2):
  - Hôpitaux Pédiatriques de Nice CHU-Lenval, Nice
  - Hôpital Armand Trousseau - APHP, Paris
- Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz, Germany
- Hungary (5):
  - Semmelweis University, 2nd Dpt of Paediatrics, Budapest
  - Heim Pál Pediatric Hospital, Budapest
  - University of Debrecen Clinical Center, Pediatric Clinic No. I., Debrecen
  - Petz Aladár County Teaching Hospital, Department of Pediatric Surgery, Győr
  - University of Pécs Clinical Centre, Pediatric Clinic, Pécs
- Romania (5):
  - Spitalul Clinic de Urgenta pentru Copii "Grigore Alexandrescu", Bucharest
  - Spitalul Clinic de Urgenta pentru Copii "Maria Sklodowska Curie", Bucharest
  - Spitalul Clinic de Urgenta pentru Copii Cluj-Napoca, Cluj-Napoca
  - Spitalul Clinic de Urgenta pentru Copii "Sfanta Maria", Iași
  - Spitalul Clinic de Urgenta pentru Copii "Louis Turcanu", Timișoara
- Serbia (4):
  - University Children' s Hospital, Belgrade
  - Mother and Child Healthcare Institute of Serbia "Dr Vukan Cupic", Belgrade
  - Clinical Centre Nis, Clinic for Pediatric Surgery and Orthopedics, Niš
  - Insititute for Health Protection of Children and Youth, Novi Sad
- Karolinska Universitetssjukhuset, Huddinge, Stockholm County, Sweden
- United Kingdom (3):
  - Birmingham Children's Hospital NHS Foundation Trust, Birmingham
  - Clesea & Westmisnter Hospital, London
  - Southampton Children's Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 18 sites in the United States, Bulgaria, France, Hungary, Romania, Serbia, and United Kingdom, from 18 January 2019 (first participant enrolled to receive the study drug) to 20 May 2022 (last participant completed).
Pre-assignment Details: Paediatric participants with excessive bleeding during surgery were randomized into 1: 1 ratio to receive Fibrin Sealant (FS) Grifols and EVICEL. A total of 197 participants were screened, out of which 186 participants were randomized (Intent-to-treat population), 178 received study treatment (modified intent-to-treat population), 171 participants completed the study.
Period: Overall Study
Arm/Group | Fibrin Sealant Grifols | EVICEL
Started | 95 | 91
Parenchymous Surgery | 46 (Participants who underwent parenchymous surgery were included.) | 43 (Participants who underwent parenchymous surgery were included.)
Soft Tissue Surgery | 45 (Participants who underwent soft tissue surgery were included.) | 44 (Participants who underwent soft tissue surgery were included.)
Safety Population (Safety population included all participants who received any amount of IP.) | 91 | 87
Completed | 87 | 84
Not Completed | 8 | 7
Not completed — Death | 1 | 2
Not completed — Consent Withdrawn by Participant | 0 | 1
Not completed — Screen Failure | 3 | 1
Not completed — Reason not Specified | 1 | 3
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all participants who were randomized, regardless of meeting intra-operative enrollment criteria and regardless of whether the IP was administered to the participant.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fibrin Sealant Grifols | EVICEL | Total
Number analyzed (Participants) | 95 | 91 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.43 (6.108) | 8.84 (6.320) | 8.63 (6.199)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 30 | 70
  Male | 55 | 61 | 116
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 11 | 24
  Not Hispanic or Latino | 82 | 80 | 162
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 86 | 89 | 175
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Hemostasis Within 4 Minutes After Treatment Start (T4)
Description: Hemostasis is defined as Grade 0 bleeding per 5-point validated bleeding severity scale (0=no bleeding and 4=Unidentified or inaccessible spurting or gush) at the target bleeding site (TBS) according to the investigator's (surgeon's) judgment, so that the surgical closure of the exposed field could begin.
Time Frame: From start of treatment until 4 minutes after treatment start (Day 1)
Population: Modified ITT (mITT) population included all participants in the ITT population who meet the intra-operative enrollment criteria, and thus treated with any amount of investigational product (IP). Overall number analyzed are the number of participants with haemostasis by 4 minutes. Number analyzed are the number of participants with parenchymous and soft tissue surgery with data available for analysis. Percentage are rounded off the single decimal point.
Measure: Number; unit: percentage of participants
Arm/Group | Fibrin Sealant Grifols | EVICEL
Number analyzed (Participants) | 91 | 87
percentage of participants
  Parenchymous Surgery: number analyzed (Participants) | 46 | 43
  Parenchymous Surgery | 100.0 | 100.0
  Soft Tissue Surgery: number analyzed (Participants) | 45 | 44
  Soft Tissue Surgery | 93.3 | 90.9
Statistical Analysis 1: Comparison: Fibrin Sealant Grifols vs EVICEL; Hemostasis by 4 Minutes (Parenchymous); Test type: Non-Inferiority — The non-inferiority was deemed to have been demonstrated if the lower limit of the 95% confidence interval (CI) exceeds 0.8; p < 0.001, Cochran-Mantel-Haenszel; Relative risk = 1, 95% CI 2-sided [0.92 to 1.09]
Statistical Analysis 2: Comparison: Fibrin Sealant Grifols vs EVICEL; Hemostasis by 4 Minutes (Soft Tissue); Test type: Non-Inferiority — The non-inferiority was deemed to have been demonstrated if the lower limit of the 95% CI exceeds 0.8; p < 0.001, Cochran-Mantel-Haenszel; Relative risk = 1.03, 95% CI 2-sided [0.91 to 1.16]

2. Secondary Outcome: Cumulative Percentage of Participants Achieving Hemostasis at the TBS by the 7 Minutes After Treatment Start (T7)
Description: Hemostasis is defined as Grade 0 bleeding at the TBS according to the investigator's (surgeon's) judgment, so that the surgical closure of the exposed field could begin. The cumulative percentage of participants achieving hemostasis at the TBS by the time points of T7 defined as an absence/cessation of bleeding (Grade 0) at the TBS by that time point without occurrence of rebleeding, Grade 3 or Grade 4 bleeding, use of alternative hemostatic treatment, and reapplication of study treatment after T4 and until TClosure.
Time Frame: From start of treatment to 7 minutes after start of treatment (Day 1)
Population: mITT population included all participants in the ITT population who meet the intra-operative enrollment criteria, and thus treated with any amount of IP. Overall number analyzed are the number of participants with haemostasis by 4 minutes. Number analyzed are the number of participants with parenchymous and soft tissue surgery with data available for analysis. Percentages are rounded off a single decimal point.
Measure: Number; unit: percentage of participants
Arm/Group | Fibrin Sealant Grifols | EVICEL
Number analyzed (Participants) | 91 | 87
percentage of participants
  Parenchymous Surgery: number analyzed (Participants) | 46 | 43
  Parenchymous Surgery | 100.0 | 100.0
  Soft Tissue Surgery: number analyzed (Participants) | 45 | 44
  Soft Tissue Surgery | 100.0 | 100.0
Statistical Analysis 1: Comparison: Fibrin Sealant Grifols vs EVICEL; Hemostasis by 7 Minutes (Parenchymous); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Relative risk = 1, 95% CI 2-sided [0.92 to 1.09]
Statistical Analysis 2: Comparison: Fibrin Sealant Grifols vs EVICEL; Hemostasis by 7 Minutes (Soft tissue); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Relative risk = 1, 95% CI 2-sided [0.92 to 1.09]

3. Secondary Outcome: Cumulative Percentage of Participants Achieving Hemostasis at the Target Bleeding Site by 10 Minutes After Treatment Start (T10)
Description: Hemostasis is defined as Grade 0 bleeding at the TBS according to the investigator's (surgeon's) judgment, so that the surgical closure of the exposed field could begin. The cumulative percentage of participants achieving hemostasis at the TBS by the time points of T10 defined as an absence/cessation of bleeding (Grade 0) at the TBS by that time point without occurrence of rebleeding, Grade 3 or Grade 4 bleeding, use of alternative hemostatic treatment, and reapplication of study treatment after T4 and until TClosure.
Time Frame: From start of treatment to 10 minutes after start of treatment (Day 1)
Population: mITT population included all participants in the ITT population who meet the intra-operative enrollment criteria and thus treated with any amount of IP. Overall number analyzed are the number of participants with haemostasis by 4 minutes. Number analyzed are the number of participants with parenchymous and soft tissue surgery with data available for analysis. Percentages are rounded off a single decimal point.
Measure: Number; unit: percentage of participants
Arm/Group | Fibrin Sealant Grifols | EVICEL
Number analyzed (Participants) | 90 | 87
percentage of participants
  Parenchymous Surgery: number analyzed (Participants) | 45 | 43
  Parenchymous Surgery | 97.8 | 100.0
  Soft Tissue Surgery: number analyzed (Participants) | 45 | 44
  Soft Tissue Surgery | 100.0 | 100.0
Statistical Analysis 1: Comparison: Fibrin Sealant Grifols vs EVICEL; Hemostasis by 10 Minutes (Parenchymous); Test type: Non-Inferiority — The non-inferiority was deemed to have been demonstrated if the lower limit of the 95% CI exceeds 0.8; p < 0.001, Cochran-Mantel-Haenszel; Relative risk = 0.98, 95% CI 2-sided [0.94 to 1.02]
Statistical Analysis 2: Comparison: Fibrin Sealant Grifols vs EVICEL; Hemostasis by 10 Minutes (Soft tissue); Test type: Non-Inferiority — The non-inferiority was deemed to have been demonstrated if the lower limit of the 95% CI exceeds 0.8; p < 0.001, Cochran-Mantel-Haenszel; Relative risk = 1, 95% CI 2-sided [0.92 to 1.09]

4. Secondary Outcome: Percentage of Participants With Treatment Failures
Description: Participants were considered treatment failures if there is a. persistent bleeding at the TBS beyond T4 b. Grade 3 or Grade 4 breakthrough bleeding from the TBS that jeopardizes participant safety according to the investigator's judgment at any moment during the 10-minute observational period and until TClosure c. Use of alternative hemostatic treatments or maneuvers (other than the study treatment) at the TBS during the 10-minute observational period and until TClosure, or use of study treatment at the TBS beyond T4 and until TClosure d. Rebleeding (Grade ≥1) at the TBS after the assessment of the primary efficacy endpoint at T4 and until TClosure.
Time Frame: From start of treatment to 10 minutes after start of treatment and until the time of completion of surgical closure (Day 1)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Fibrin Sealant Grifols | EVICEL
Number analyzed (Participants) | 91 | 87
percentage of participants
  Parenchymous Surgery: number analyzed (Participants) | 46 | 43
  Parenchymous Surgery | 0 | 0
  Soft Tissue Surgery: number analyzed (Participants) | 45 | 44
  Soft Tissue Surgery | 0 | 0

ADVERSE EVENTS:
Time Frame: From signing informed consent form up to 7 days post study completion (Up to approximately 47 days)
Description: Safety population included all participants who received any amount of IP.
Arm/Group | Fibrin Sealant Grifols | EVICEL
All-Cause Mortality (participants affected / at risk) | 1/91 | 2/87
Serious Adverse Events (participants affected / at risk) | 8/91 | 9/87
Other Adverse Events (participants affected / at risk) | 20/91 | 13/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fibrin Sealant Grifols (N=91) | EVICEL (N=87)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Transaminases increased (Investigations) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Intussusception (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fibrin Sealant Grifols (N=91) | EVICEL (N=87)
Hypertension (Vascular disorders) | 2 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0
Mechanical ventilation complication (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 0
Blood magnesium decreased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 1
Oxygen saturation decreased (Investigations) | 1 | 0
Platelet count increased (Investigations) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 3
Generalised oedema (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 5
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 5 | 3
Acquired hydrocele (Reproductive system and breast disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Postoperative abscess (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the Study, after providing Sponsor thirty days' notice prior to submitting a manuscript or other materials related to the Study to any outside party. At Sponsors' request, Site will remove any Confidential Information (other than Study results), and Site will upon Sponsors' request, delay publication or presentation for a period of up to one hundred twenty days to allow Sponsor to protect its interests in any Sponsor Inventions.

DOCUMENTS (2):
  • Study Protocol (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/06/NCT03461406/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/06/NCT03461406/SAP_001.pdf